CLINICAL TRIAL: NCT06389669
Title: Low Flow Anaesthesia is Good But Feasible?
Brief Title: Is Low Flow Anaesthesia Feasible?
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Yusuf Ziya ÇOLAK, Associate Professor, MD, Inonu University
Other Study IDs: Inonu LTI
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia
Keywords: Low Flow Anaesthesia; Closed-Circuit Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although low-flow anaesthesia (LFA) has been described for many years and its benefits are known, its clinical use has been limited. Concerns about the risk of hypoxia contributed to this situation. Although the risk of hypoxia is almost prevented with advanced anaesthesia machines, the use of LFA has not reached the desired levels. However, in recent years, as adverse developments related to climate change have started to affect us all, LFA has started to be on the agenda of anaesthetists again. In this study, our aim is to examine the feasibility of its clinical use in order to popularise the use of LFA.

DETAILED DESCRIPTION:
ASA 1-2 patients who will undergo elective surgery under general anaesthesia in 38 operating rooms of Inonu University Faculty of Medicine will be prospectively recruited for 3 months (May-June-July). Emergency cases, patients under the age of 18 and over 65, laparoscopic surgeries, heart-lung surgeries that may impair oxygenation will not be included in the study.

Inhaler anaesthesia will be administered after anaesthesia induction and tracheal intubation. Fresh gas flow (FGF) will be determined as 1 l/min, MAC=1, FiO2=40% with target controlled automatic gas control mode (AGC). FGF will be decreased to 0.5 l/min 10 minutes after surgical incision, if successful, it will be decreased to 0.3 l/min 10 minutes later and it will be checked whether it is successful. The study will be terminated and FGF will be increased to 1 l/min again.

Demographic data of the patients and FGF levels that can provide FiO2=40% will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery under general anaesthesia

Exclusion Criteria:

* Emergency operations
* Previously diagnosed heart, lung, liver and kidney disease
* Surgeries that may impair oxygenation (laparoscopic, Heart, Lung surgeries)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA 1-2 patients who will undergo elective surgery under general anaesthesia in 38 operating rooms of Inonu University Faculty of Medicine will be prospectively recruited for 3 months (May-June-July). Emergency cases, patients under the age of 18 and over 65, laparoscopic surgeries, heart-lung surgeries that may impair oxygenation will not be included in the study.
Sampling Method: Probability Sample
Enrollment: 785 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Feasibility of Low Flow Anaesthesia | The measurement will start 10 minutes after the surgical incision and end 20 minutes later
  To determine the lowest amount of fresh gas flow, most suitable for the patient and, which can provide FiO2=40% level

SECONDARY OUTCOMES:
Factors affecting oxygen consumption | The measurement will start 10 minutes after the surgical incision and end 20 minutes later
  To find out which of the patient's physical characteristics that affect oxygen consumption may be determinant.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Z Colak, Assoc.Prof., Principal Investigator — Inonu University Anaesthesiology and Reanimation Department
Locations (1):
- Inonu Univercity, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided